CLINICAL TRIAL: NCT06175767
Title: A Phase IIa, Randomized, Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of MT101-5 in Subjects with Early Parkinson's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of MT101-5 in Subjects with Early Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mthera Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MT101-PD-002
Record Dates: First submitted 2023-11-22; First posted 2023-12-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Screening Phase (Day -28 to Day -1, up to 28 days): (Experimental): Screening phase is designed to determine subject's eligibility to proceed to Randomization and the Treatment Phase of the study. During this phase, a series of assessments will be performed to determine subject eligibility as per inclusion and exclusion criteria.
  Subjects who meet eligibility criteria, but have some abnormal laboratory values, based on PI review a repeat laboratory sample may be collected. The repeat laboratory reports should be reviewed by the PI to confirm eligibility prior to randomization.
  Subjects who fail to meet eligibility criteria during the Screening phase will be considered screen failures and will be exited from the study. Subjects who meet the eligibility criteria will be scheduled for randomization visit.
  Interventions: Drug: MT101-5
- Randomization and Double-Blind Treatment Phase (TV0- TV3, 12 weeks): (Experimental): Subjects who have successfully completed the Screening phase will enter the Randomization and Double-Blind treatment phase of the study. Subjects will take the assigned randomized treatment, MT101-5 at 400 mg, 600 mg or placebo for 12 weeks. MT101-5 and matching placebo are oral tablets that will be taken as six tablets two times a day (b.i.d.) at least 2 hours before or 2 hours after meal in the morning and evening daily during this study.
  Interventions: Drug: MT101-5
- Follow-up Phase (FUV, 4 weeks ± 3 days) (Experimental): The follow-up phase will consist of a follow-up visit at the end of the Double-Blind Treatment phase.
  Interventions: Drug: MT101-5

INTERVENTIONS:
Drug: MT101-5 — Tablet

SUMMARY:
A Phase IIa, Randomized, Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of MT101-5 in Subjects with Early Parkinson's Disease. Primary objective of the study is to evaluate the safety and tolerability of MT101-5 400 mg and 600 mg oral tablet total daily dose compared to Placebo in subjects with Parkinson's Disease.

DETAILED DESCRIPTION:
The study will include three phases: a 4-week Screening Phase, a 12-week Double-Blind Treatment Phase, and a 4-week Follow-up Phase.

Screening Phase (Day -28 to Day -1, up to 28 days):

Screening phase is designed to determine subject's eligibility to proceed to Randomization and the Treatment Phase of the study. During this phase, a series of assessments will be performed to determine subject eligibility as per inclusion and exclusion criteria.

At the Screening Visit, prior to any study-related procedures, a written informed consent will be obtained from the subject by the Investigator or suitable qualified personnel. Screening procedures will be conducted per the study schedule of events. All screening information will be documented in the case report forms.

Subjects who meet eligibility criteria, but have some abnormal laboratory values, based on PI review a repeat laboratory sample may be collected. The repeat laboratory reports should be reviewed by the PI to confirm eligibility prior to randomization.

Subjects who fail to meet eligibility criteria during the Screening phase will be considered screen failures and will be exited from the study. Subjects who meet the eligibility criteria will be scheduled for randomization visit.

Randomization and Double-Blind Treatment Phase (TV0- TV3, 12 weeks):

Subjects who have successfully completed the Screening phase will enter the Randomization and Double-Blind treatment phase of the study. Subjects will take the assigned randomized treatment, MT101-5 at 400 mg, 600 mg or placebo for 12 weeks. MT101-5 and matching placebo are oral tablets that will be taken as six tablets two times a day (b.i.d.) at least 2 hours before or 2 hours after meal in the morning and evening daily during this study.

Randomization/Treatment Visit 0 (TV0):

On Day 0 prior to randomization, the subject's continued eligibility will be evaluated. Subjects who continue to be eligible will be randomized in a 1:1:1 ratio to one of the following treatment groups and assigned the study treatment kit:

* Group 1: MT101-5 400 mg divided b.i.d. (Total daily dose of 400 mg, combination of four 50 mg MT101-5 tablets and two placebo tablets, taken as six tablets two times daily at least 2 hours before or 2 hours after meal).
* Group 2: MT101-5 600 mg divided b.i.d. (Total daily dose of 600 mg, 50 mg tablets taken as six tablets two times daily at least 2 hours before or 2 hours after meal).
* Group 3: Placebo tablet (0 mg MT101-5) divided b.i.d. (Total daily dose of 0 mg, 0 mg taken as six placebo tablets two times daily at least 2 hours before or 2 hours after meal).

Treatment Visits 1 (TV1) through 3 (TV3):

Clinic treatment visits TV1 through TV3 will be conducted every four (4) weeks (± window periods). During each of these visits, study evaluations will be conducted per the study schedule of events and sufficient supply of MT101-5 or placebo till the next treatment visit will be dispensed.

Treatment Visit 3 (TV3) will be the end of treatment (EOT) clinic visit. Study evaluations, review of the adverse events, concomitant medications and final study treatment accountability will be conducted.

Follow-up Phase (FUV, 4 weeks ± 3 days)

The follow-up phase will consist of a follow-up visit at the end of the Double-Blind Treatment phase.

ELIGIBILITY:
Inclusion Criteria

Subjects will be eligible for enrollment in the study only if they meet ALL of the following criteria:

1. Male or female subjects who are between 30 and 79 years old inclusive with a clinical diagnosis of Parkinson's disease as per UK Brain Bank Criteria for two (2) years or less at screening.
2. Hoehn and Yahr I or II at screening.
3. Subjects who are newly diagnosed & currently not on any Parkinson's disease medication (or) subjects who are on stable doses for at least 4 weeks prior to screening on Amantadine or anticholinergics for treatment of Parkinson's disease (1) Note: Subjects that had anti-parkinsonian medication (including levodopa, dopamine agonists, entacapone and monoamine oxidase-B inhibitors) discontinued at least 60 days prior to screening, e.g., for intolerance, may be considered eligible if all other eligibility requirements are met.
4. Without clinically significant abnormalities in physical exam, neurological exam and laboratory assessments (urine/blood routine, biochemical tests and ECG) which would exclude the subject from the study in the opinion of the Investigator. For aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) the screening levels should be ≤ 2 times upper limit normal.
5. Subject is capable of providing informed consent and is willing to sign the ICF prior to study Screening and agrees to comply with the study protocol requirements.

Exclusion Criteria

Subjects will be eligible for enrollment in the study only if they meet NONE of the following criteria:

1. Subject has an atypical parkinsonian syndrome or secondary parkinsonism (e.g., due to drugs, metabolic neurogenetic disorders, encephalitis, cerebrovascular disease or degenerative disease).
2. Subjects with history of neurosurgical intervention for Parkinson's disease.
3. Subjects who meet the DSM-V criteria at screening for bipolar disorder, major depressive disorder, psychotic disorders, or any other comorbid mental disorders that in the opinion of the Investigator may interfere with study conduct and results interpretation.
4. Subjects with clinical diagnosis of dementia (MMSE score <24) as determined by the investigator using Mini-Mental State Examination (MMSE).
5. Female subjects who are pregnant or breast feeding.
6. Initiation of any anti-parkinsonian medication (including levodopa, dopamine agonists, entacapone and monoamine oxidase-B inhibitors) for the duration of the trial.
7. Initiation of Amantadine or anticholinergics for newly diagnosed subjects or change in the dosage of Amantadine or anticholinergics during the trial for subjects who were on stable doses for 4 weeks prior to screening.
8. Medical or recreational use of marijuana or THC-containing compounds within 3 months of screening visit and for the duration of the trial.
9. Subjects who used investigational drugs or devices within 60 days prior to screening or investigational biologics within the last 6 months prior to screening.
10. Subjects with a clinically significant medical or surgical condition, including major surgeries within 28 days prior to enrollment.
11. The subject has a known allergy or hypersensitivity to any component of the formulation.
12. The subject has a history of alcohol abuse (defined as an alcohol intake more than 21 units per week) or a history of drug abuse within the 6 months before study drug administration, or a history of substance abuse deemed significant by the investigator. A unit of alcohol is defined as 240 mL of beer, 120 mL of wine, or 1 single shot of spirits.
13. Women of child-bearing age who are sexually active but decline to take proper contraceptive measures during the study period

Note: To be eligible for the study, Women of childbearing potential (WOCBP) and Women not of childbearing potential are eligible to participate. Both women of childbearing potential and women of no childbearing potential should use an approved method of birth control and agrees to continue to use this method for the duration of the study (and for 30 days after taking the last dose of investigational product).

Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile or 2 years post-menopausal. All male subjects/partners of WOCBP must agree to consistently and correctly use a condom for the duration of the study and for 30 days after taking the study drug. In addition, subjects may not donate ova or donate sperm for the duration of the study and for 30 days after taking the last dose investigational product.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-14 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Change from baseline to week 12 after the first study drug administration
  An adverse event (AE) is defined as any unfavorable or unintended sign, symptom, or disease that occurs or is reported by the patient to have occurred, or a worsening of a pre-existing condition. An adverse event may or may not be related to the study treatment.
Incidence of withdrawals due to Adverse Events (AEs) | Change from baseline to week 12 after the first study drug administration
  Incidence of withdrawals due to Adverse Events (AEs) defined above
Incidence of serious adverse events (SAEs) | Change from baseline to week 12 after the first study drug administration
  Adverse event that results in death, is life threatening, Requires subject hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Change from baseline to week 12 after the first study drug administration
  Suicidal ideation/suicidal behavior assessment tool. Score ranges from 2 to 25, with the higher number indicating more intense ideation.
Change of blood pressure (both systolic and diastolic blood pressures) | Change from baseline to week 12 after the first study drug administration
Change of body temperature | Change from baseline to week 12 after the first study drug administration
Change of respiratory rate | Change from baseline to week 12 after the first study drug administration
ECG ventricular rate (beats per minute) | Change from baseline to week 12 after the first study drug administration
ECG PR interval (msec) | Change from baseline to week 12 after the first study drug administration
ECG QRS interval (msec) | Change from baseline to week 12 after the first study drug administration
ECG QT interval (msec) | Change from baseline to week 12 after the first study drug administration
ECG QTc interval (msec) | Change from baseline to week 12 after the first study drug administration

SECONDARY OUTCOMES:
Movement Disorder Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) total score | Change from baseline to week 12 after the first study drug administration
  A multimodal scale assessing both impairment and disability. Score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability
Schwab and England (S&E) Scale total score | Change from baseline to week 12 after the first study drug administration
  Scale that reflects the speed, ease, and independence with which an individual performs daily activities. Score range from 0% to 100%. Higher the percentage better the outcome.
Parkinson's Disease Questionnaire (PDQ-39) total score | Change from baseline to week 12 after the first study drug administration
  Patient reported rating scale in Parkinson's disease. Score between 0 and 100. Lower scores reflect better quality of life.
Hoehn and Yahr (H&Y) scale total score | Change from baseline to week 12 after the first study drug administration
  System for describing how the symptoms of Parkinson's disease progress. Score range from 0 to 5. Higher the score worse the outcome.
Clinical Global Impression-Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I) scale score. | Change from baseline to week 12 after the first study drug administration
  The CGI measures global severity of illness at a given point in time. Score range from 1 to 7. Higher the score worse the outcome.

OTHER OUTCOMES:
Change from baseline of CSF levels of alpha-synuclein | Change from baseline to week 12 after the first study drug administration
  Analysis to determine CSF concentrations of alpha-synuclein
Discovery of biomarkers for MT101-5 as significant DEPs (differentially expressed proteins) with >2-fold change between MT101 and PD patient groups. | Change from baseline to week 12 after the first study drug administration
  The protein identification and expression of the CSF sample